CLINICAL TRIAL: NCT03353363
Title: A Comparison of Post-Incisional Wound Infiltration of Liposomal Bupivacaine to Plain Bupivacaine for Post-Operative Pain Control in Elective Cesarean Delivery: A Randomized Double Blind Placebo Controlled Trial
Brief Title: Wound Infiltration of Liposomal Bupivacaine v Plain Bupivacaine for Post-Op Pain Control in Elective Cesarean Delivery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Brian M. Fitzgerald, MD, Staff Anesthesiologist, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C.2017.156
Record Dates: First submitted 2017-11-16; First posted 2017-11-27 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2017-11

CONDITIONS: Bupivacaine; Pain, Postoperative
Keywords: cesarean delivery; liposomal bupivacaine; Exparel; bupivacaine; wound infiltration
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-Blind Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Normal Saline (Placebo Comparator): Subject will receive 20ml of normal saline infiltration
  Interventions: Drug: Placebos
- Plain Bupivacaine (Experimental): Subject will receive 20ml of 0.5% plain bupivacaine infiltration (100mg)
  Interventions: Drug: Bupivacaine
- Liposomal Bupivacaine (Experimental): Subject will receive 20ml of liposomal bupivacaine infiltration (266mg) non-expanded
  Interventions: Drug: Liposomal bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — After patients receive their spinal anesthetic and as the Pfannenstiel incision is being closed, an equal volume (20ml, administered via two 10ml syringes) of bupivacaine 0.5% plain will be infiltrated into the wound by the obstetrician team in a standardized fashion.
  Arms: Plain Bupivacaine
Drug: Liposomal bupivacaine — After patients receive their spinal anesthetic and as the Pfannenstiel incision is being closed, an equal volume (20ml, administered via two 10ml syringes) of one liposomal bupivacaine will be infiltrated into the wound by the obstetrician team in a standardized fashion.
  Other Names: Exparel
  Arms: Liposomal Bupivacaine
Drug: Placebos — After patients receive their spinal anesthetic and as the Pfannenstiel incision is being closed, an equal volume (20ml, administered via two 10ml syringes) of normal saline will be infiltrated into the wound by the obstetrician team in a standardized fashion.
  Arms: Normal Saline

SUMMARY:
Randomized double blind placebo controlled trial to compare the post-operative pain control advantages of post-incisional wound infiltration with liposomal bupivacaine to plain bupivacaine in patients presenting for elective caesarean delivery.

DETAILED DESCRIPTION:
Participants will include women with uncomplicated singleton pregnancies, ≥37 weeks gestation, ≥18 years old presenting and presenting for elective caesarean delivery with a planned spinal anesthetic with a standardized amount of intrathecal morphine (ITM). Exclusion criteria include patients: not receiving a spinal anesthetic, receiving a spinal anesthetic that required supplemental intraoperative pain medications (ketamine, epidural narcotics, intravenous narcotics, etc), on chronic opioids, American Society of Anesthesiologist (ASA) physical status class III or higher (Note: An ASA I patient is defined as a normal healthy patient, an ASA II patient is defined as a patient with mild systemic disease and any patient that with severe systemic disease or a disease that is incapacitating would be classified as an ASA III or higher) or those that have known hypersensitivity to bupivacaine hydrochloride, amide-type local anesthetics, or any component of the formation, and any subject with hepatic or renal impairment.

A three-arm study will be used: (a) control group (placebo of normal saline) (b) plain bupivacaine group and (c) liposomal bupivacaine group. After patients receive their spinal anesthetic and as the Pfannenstiel incision is being closed, an equal volume (20ml, administered via two 10ml syringes) of one of the three solutions will be infiltrated into the wound by the obstetrician team in a standardized fashion.

ELIGIBILITY:
Inclusion Criteria:

1. ASA I or II women with uncomplicated singleton pregnancies
2. ≥37 weeks gestation
3. ≥18 years old presenting
4. Presenting for elective caesarean delivery with a planned spinal anesthetic with a standardized amount of intrathecal morphine (ITM).
5. Able to provide informed consent.

Exclusion Criteria:

1. Subject is not a candidate for a spinal anesthetic
2. Subject receives a spinal anesthetic that required supplemental intraoperative pain medications (ketamine, epidural local anesthetic, epidural narcotics, intravenous narcotics, etc)
3. Subject is on chronic opioids.
4. Subject is an ASA class III or higher.
5. Subject has a known hypersensitivity to bupivacaine hydrochloride, amide-type local anesthetics, or any component of the formation,
6. Subject has hepatic or renal impairment that is concerning, as determined by the surgeon or anesthesiologist.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants will include ASA I or II women with uncomplicated singleton pregnancies, ≥37 weeks gestation, ≥18 years old presenting and presenting for elective caesarean delivery
Enrollment: 132 (Estimated)
Dates: Start 2017-10-18 (Actual); Primary Completion 2018-10-18 (Estimated); Study Completion 2019-02-18 (Estimated)

PRIMARY OUTCOMES:
Post-operative Analgesia | Thru 24 hours
  VAS pain intensity scores (at rest)
Post-operative Analgesia | Thru 48 hours
  VAS pain intensity scores (at rest)

SECONDARY OUTCOMES:
Opioid use in the post-operative period | Thru 72 hours
  Post-operative opioid consumption
Length of Stay (LOS) | Thru 72 hours
  Reduction in LOS
Time to first ambulation | Thru 72 hours
  Time to ambulation
Breast feeding initiation | Thru 72 hours
  Time to breast feeding initiation
Sole breastfeeding | Thru 72 hours
  Percentage of subjects solely breastfeeding at the time of discharge
Increased operative time | Thru 72 hours
  Increased operative time for cesarean delivery
Pain control at 2 hours post-cesarean delivery | Thru 2 hours
  VAS pain intensity at 2 hours
Wound Complication | 14days post-operatively
  Wound complication

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Fitzgerald, MD, Principal Investigator — Brooke Army Medical Center
Locations (1):
- Brooke Army Medical Center, Fort Sam Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: By request.
Access Criteria: By request.